CLINICAL TRIAL: NCT04695730
Title: Comparison Between Two Physical Therapy Treatments in Patients With Nonspecific Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Paolo Pillastrini, Professor, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 679/2020/Sper/AOUBo
Record Dates: First submitted 2020-12-13; First posted 2021-01-05 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Non-specific Chronic Neck Pain
Keywords: neck pain; chronic neck pain; musculoskeletal disorder
MeSH Terms: conditions — Neck Pain; Musculoskeletal Diseases | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Masking Description: Statistician (data analyst) will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active physical therapy (Active Comparator): Active intervention (including both pain education and home exercises). A 60-minutes education session will be provided, concerning pain mechanisms and management and a demonstration of the exercises to perform individually at home. Home exercises will be performed daily. To support patients during the treatment, a booklet will be created. One 30-minutes booster session will be planned after 4 weeks. Patients will follow this active intervention for 8 weeks.
  Interventions: Other: Active physical therapy (including both pain education and home exercises)
- Active physical therapy plus manual therapy (Experimental): Participants in the Group 2 will receive active intervention plus 8 "Pompage" technique sessions (1 session/week). In these sessions (30 minutes each), "Pompage" technique will be performed by a physical therapist.
  Interventions: Other: Active physical therapy plus manual therapy

INTERVENTIONS:
Other: Active physical therapy (including both pain education and home exercises) — One session (60 minutes). In this session, a physical therapist will explain and demonstrate the exercises to perform individually at home. Exercises will be performed daily. In addition, an education session will be provided, concerning pain mechanisms and management. To support patients during the treatment, a booklet will be created.
  One booster session (30minutes) will be planned after 4 weeks. Patients will follow the active treatment for 8 weeks.
  Arms: Active physical therapy
Other: Active physical therapy plus manual therapy — Participants in the Group 2 will receive active intervention plus 8 "Pompage" technique sessions (1 session/week). In these sessions (30 minutes each), "Pompage" technique will be performed by a physical therapist.
  Arms: Active physical therapy plus manual therapy

SUMMARY:
Introduction: Non-specific chronic neck pain is a very prevalent condition in the population ranging from 45% to 54%. Several conservative treatments have been shown to be effective and are currently used in clinical practice. However, among the physical therapy ones, no study evaluated the effectiveness of Pompage techniques in addition to an active treatment.

This protocol describes a controlled, randomized trial that aims to assess the effectiveness of two physical therapy treatments in patients with chronic non-specific neck pain.

Methods: Seventy subjects with chronic nonspecific neck pain from 18 to 80 years will be recruited according to the inclusion criteria.

Afterwards they will be randomized to one of the 2 groups: group 1 (G1) will undergo an active intervention and group 2 (G2) will receive the same active intervention plus manual technique. Active intervention, according to the current guidelines on non-specific neck pain, will be a treatment including both pain education and home exercises; manual technique will be the so-called "Pompage" technique.

A booster session will be planned for both groups after 4 weeks from the beginning of the trial, to reinforce the patients adherence to the self-treatment.

The patients will be evaluated before the treatments (baseline, T0), after 8 weeks from the beginning of the treatments (T1), and 6 months after the end of the treatments (T2).

The primary outcome will be pain perception, which will be assessed using a Visual Analogue Scale (VAS).

The secondary outcomes will be: kinesiophobia (measured with the Tampa Scale of Kinesiophobia - TSK), physical function (measured with the Neck Disability Index - NDI), active cervical range of motion - ROM (measured with the "CROM Deluxe" device), patient satisfaction for treatment (measured with the Physical Therapy Satisfaction Questionnaire - PTPSQI(15)), and subjective perception of improvement (measured with the Global Perceived Effect - GPE).

Adverse effects will be registered. Discussion: Considering that there is no consensus on the use of Pompage techniques in addition to an active treatment in individuals with nonspecific chronic neck pain, our protocol will be the basis for the use of these techniques by health professionals and for new studies to be performed.

DETAILED DESCRIPTION:
PROTOCOL OF INTERVENTIONS

The intervention of group 1 (G1) is based on education and selective strengthening exercises for cervical muscles, and involves a protocol that must be performed by the patient for 8 weeks. Halfway through the course (at the end of the fourth week) the physical therapist will carry out a reinforcement session, to monitor the clinical situation, motivate the patient and resolve any doubts (booster session).

In group 2 (G2) the "Pompage" treatment will be added to this intervention.

HOME EXERCISES: CONTENTS

In the first session supervised by a physical therapist, lasting 30 minutes, the patient will be taught all the home exercises that he/she will have to perform and will be given:

1. a hard copy with the exercise reminder;
2. a diary for recording the daily execution of the exercises. The patients will be instructed to perform the exercises on a daily basis, without feeling pain. These exercises focus on strengthening the deep muscles of the neck; cranio-cervical flexor muscles and cervical extensors.

PAIN EDUCATION: CONTENTS

The educational intervention will take place verbally in a 30-minute session (explanation by the physical therapist), and will be supported by images, diagrams and summaries.

During this intervention, the patient will be provided with information on chronic non-specific cervical pain and on "pain neuroscience education". The education session will focus on explaining the mechanisms through which the body perceives and interprets pain. The aim is to make the patient aware that experiencing pain does not necessarily mean that there is a damage on a part of the body. During this educational session, the physical therapist will try to encourage the patient to ask questions.

At the end of this session, the patient will be given an information booklet on pain, with references to the themes just explored. This booklet provides further examples and ideas for elaborating and fixing the concepts learned during the session supervised by the physical therapist.

MANUAL THERAPY: CONTENTS

The treatment of group 2 (G2) combines the previous treatments with eight 30-minutes sessions of passive manual therapy, using the "Pompage" technique, carried out according to the indications shown in the monograph: "Zanella F, Vanti C. Pompage technique. The myofascial release. Piccin, Padua, 2015." The "Pompage" technique includes gradual and progressive soft tissue and fascia mobilization procedures, with the aim to obtain the myofascial release. This procedure is performed without provoking pain or forcing movements beyond the passive physiological range of motion. It consists of an alternation of rhythmic pressure and decompression, located at cervical joints and muscles (e.g. Trapezius Superior, Levator scapulae, Scalenus, Sterno-Cleido-Occipito-Mastoideus, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Female and male subjects aged between 18 and 80 years with non-specific neck pain lasting for more than 3 months.
* Informed consent

Exclusion Criteria:

* Subjects with acute or subacute neck pain;
* Subjects with specific etiology for neck pain (e.g. trauma, herniated disc, vertebral deformities, fractures);
* Subjects with central or peripheral neurological signs;
* Individuals with systemic diseases, neuromuscular diseases, rheumatic diseases, cognitive deficit, tumors;
* Subjects who underwent surgery within 6 months preceding enrollment;
* Subjects who underwent physical therapy treatment within 6 months preceding enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Changes in neck pain | At baseline, 8 weeks, and 6 months.
  Visual Analogue Scale (VAS). VAS is a unidimensional measure of pain intensity. The scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]).

SECONDARY OUTCOMES:
Changes in neck disability | At baseline, 8 weeks, and 6 months.
  Italian version of Neck Disability Index (NDI) The test can be interpreted as a raw score, with a maximum score of 50, or as a percentage and includes a total of 10 items.
  Score: /50 Transform to percentage score x 100 = %points
Changes in Kinesiophobia/Fear of movement | At baseline, 8 weeks, and 6 months.
  Italian version of Tampa Scale of Kinesiophobia (TSK). Tampa Scale of Kinesiophobia (TSK), provides a measure of fear of movement or injury. The Italian version comprises 13 item divided in two subscales: TSK 1 - Activity Avoidance, and TSK 2-Harm.
  * TSK 1 - Activity Avoidance (item 1, 2, 10, 14, 15, 17):___/24
  * TSK 2 - Harm (item 3, 5, 6, 7, 9, 11, 13):___/28 The maximum score is 52. An higher score is related to an higher level of fear.
Changes in Active Cervical Range of Motion | At baseline, 8 weeks, and 6 months.
  "CROM Deluxe" device
Assessment of the satisfaction for physical therapy | At 8 weeks and 6 months.
  Italian version of Physical Therapy Satisfaction Questionnaire - (PTPSQ-I(15) PTPSQ-I(15) consists of 15 items; for each item the score ranges from 1 to 5. An higher score is related to an higher level of satisfaction.
Assessment of the global perception of improvement on a 7-points Likert Scale | At 8 weeks and 6 months.
  Global Perceived Effect (GPE) questionnaire. The GPE is composed of 1 question on a 7-point Likert-type scale evaluating the subjective self-reported improvement or deterioration after the intervention. GPE is widely used in the physical therapy literature. On the basis of GPE score, patients will be dicotomized into "improved" (a score of 1-3 on the GPE) and "worsened" (a score of 5-7 on the GPE).

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Pillastrini, Professor, Principal Investigator — University of Bologna
Locations (1):
- University of Bologna - Italy, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No